

The Effect of School Lunch
Program (SLP) Towards
Nutrition Knowledge, Attitude,
Practices and Nutrition Status of
Adolescents in Islamic Boarding
School

Cooperation
Department of Community Nutrition
Faculty of Human Ecology, IPB
PT. AJINOMOTO Indonesia

December 18 2017

# **Informed Consent to Obtain Respondent Approval**

### "School Lunch Program

## FOR THE STUDENTS OF DARUSSALAM ISLAMIC BOARDING SCHOOL"

#### Willingness to participate

We are inviting you to participate in this activity. The following information is provided to help you make a decision about whether you wish to participate or not. If there is something unclear and you want to ask a question, please do so directly.

#### **Basis for the selection of respondents**

You were chosen as a respondent because you are a student of the Darussalam Islamic Boarding School and are currently staying at the Islamic Boarding School, and do not suffer from chronic illness with BMI for age <-3 SD and severe anemia.

#### Study objectives

The general objective of this activity is to provide nutritional education and lunch for students in an effort to improve knowledge and attitudes towards a balanced diet, clean and healthy behaviors well as, improve nutritional status, decrease anemia, as well as learning ability / academic achievement. In particular this activity aims to:

- 1. Improve student knowledge regarding balanced diet.
- 2. Improve students' attitude towards clean and healthy living.
- 3. Increase energy and nutrient intake and the quality of student food consumption
- 4. Improve nutritional status
- 5. Increase hemoglobin levels (decrease anemia status) in students
- 6. Improve students' physical fitness.
- 7. Increase student's concentration (instantaneous memory)
- 8. Increase student attendance in learning activities at school

#### **Research procedure**

You will be asked to participate in a class that relates to nutritional education and consume the food served as lunch consisting of a complete menu consisting of rice, animal or/and vegetable protein sources, vegetables and fruit to be provided to you for 2 semesters. Prior to this activity, we will take a blood sample (10 microliters; to analyze hemoglobin levels). A doctor will take the blood sample and carry out a medical examination. At the middle and end of the activity, another blood sample will be taken and a medical examination carried out in order to assess the benefits.

Apart from that, you will also be asked some questions using questionnaires / interview guides. Questions include students' economic social, daily food consumption, nutritional status, knowledge regarding a balanced diet and clean and healthy living practices.

#### Possible risk

There are no potential risks associated with the implementation of this program. The food provided for consumption for 2 semesters is the food that is usually consumed because it uses local food obtained from the market around the Islamic Boarding School and is processed and served by the canteen team at the Islamic Boarding School who have been trained by the team on this program.

#### **DISCONTINUATION OF THE STUDY**

You will be invited to withdraw from the study if there is any suspect that he/she is not following the instructions. If the subjects want, for personal reason, to withdraw from the study, he/she will be free to do so, after having informed the experimenter.

The study will be discontinued should any adverse effect due to the treatment be reported. At present there is no clue to suspect any adverse effect. The subject will be discontinued if he/she experience vomiting during the treatment period.

#### **Decision to Participate**

The decision to participate or not is entirely your choice, there is no coercion (**voluntary**).

#### **Incentive**

None

#### **Compensation for participation**

You will be given nutritional education and lunch to be consumed every day for 2 semesters and get balanced nutrition education and clean and healthy lifestyle behavior throughout the program.

#### Special conditions

In the event of any complaints or disruptions related to this program during the program period, you can immediately contact the team directly, or using the contact number stated at the end of the script *informed consent* 

#### **Confidentiality guarantee**

All information obtained from this activity will be kept confidential. The information collected will be presented in a scientific forum, but your identity will be kept secret.

#### **Ethical considerations**

This study will be conducted in accordance with the Declaration of Helsinki (http://www.wma.net/en/30publications/10policies/b3/) and Ethical Guidelines for Medical and Health Research Involving Human Subjects (http://10.136.68.34/keijiban/K242/Ethical%20Guidelines%20for%20Medical%20 anf%20Health%20Research%20Involving%20Human%20Subjects.pdf).

Procedures are fully explained to all subjects, and written informed consent is obtained. This study protocol will be conducted after approval by the Clinical Research Ethics Committee of Bogor University and Ajinomoto Co., Inc.

At any time, the volunteer (or his/her legal representative) may withdraw from the study. Should this happen, the partial data will be deleted. The waiver operated by the subject (or his/her legal representative) will not have any consequence on any other treatment that the subject should need, which will be provided according to the best practices. If the new information about the test during the test has been obtained, the consent again been providing information.

#### **Rights of respondents**

We have already explained your rights as a respondent. If you still have questions, contact Dr. Rimbawan at the activity secretariat by calling 0251 (621363).

#### Willingness to participate and / or resign

You are free to decide not to participate in this activity, or to resign, **without** any sanctions. We hope that your decision to resign will not affect the relationship between the team and the Islamic Boarding School.

Thank you for your kind attention.

# LETTER OF AGREEMENT TO PARTICIPATE IN THE "School Lunch Program FOR STUDENTS OF THE DARUSSALAM ISLAMIC BOARDING SCHOOL"

.

After receiving an explanation of the objectives, procedures, possible benefits and risks and answers to my questions provided by the School Lunch Program Team for the students of Darussalam Islamic Boarding School, I

Name

| Age | : | |
|---|---|---|
| Class | : | |
| Hereby state with full awa | reness, that I am r | ready to participate, be interviewed |
| and undergo a medical exa | mination (physical | and biochemical) as a subject in the |
| "SCHOOL LUNCH PRO | GRAM FOR THE | STUDENTS OF DARUSSALAM |
| ISLAMIC BOARDING SO | CHOOL" from start | to finish; noting that all data abou |
| me will be kept confidential and if, at any time during my research period, I am | | |
| harmed in any way due to | this program I have | e the right to cancel this agreement |
| without being subject to a | ny sanctions. | |
| 1 | Bogor, | 2017 |
| The one making the stater | nent | |
| Student ( | | ) |
| ( | | ) |
| I as narent/ legal guardia | n of the student he | ereby state with full awareness, tha |
| he/she is approved to part | | • |
| Parent/ legal guardian | | |
| ( | | ) |
| Management | Witness of the Darussalam 1 | Islamic Boarding School |
| Hanagement | or the Darassalam i | islamic boarding school |
| ( | | ) |